CLINICAL TRIAL: NCT05961592
Title: A Single and Repeat Dosing Study of the Safety, Drug Exposure and Clinical Activity of R-2487 in Patients With Rheumatoid Arthritis
Brief Title: R-2487 in Patients With Rheumatoid Arthritis
Acronym: R-2487-RA01
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Rise Therapeutics LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RISE-2487-RA01
Record Dates: First submitted 2023-07-18; First posted 2023-07-27 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-08

CONDITIONS: Arthritis, Rheumatoid
Keywords: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Pharmaceutical Preparations

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Four (4) week open label dose for Rheumatoid Arthritis patients (Experimental): R-2487 DP administered daily for 28 days
  Interventions: Drug: R-2487 DP
- Six (6) week open label dose for Rheumatoid Arthritis patients (Experimental): R-2487 DP administered daily for 42 days
  Interventions: Drug: R-2487 DP
- Four (4) week open label dose for Rheumatoid Arthritis with Secondary Sjorgrens Syndrome patients (Experimental): R-2487 DP administered daily for 28 days
  Interventions: Drug: R-2487 DP

INTERVENTIONS:
Drug: R-2487 DP — Probiotic
  Other Names: Drug

SUMMARY:
The goal of this study is to determine the safety and tolerability of orally taken probiotic (R-2487) in patients with Rheumatoid Arthritis.

Patients will take an oral dosage of probiotic (R-2487) and physicians will assess and measure their Rheumatoid Arthritis. Blood and fecal evaluations of inflammation and assessment of probiotic (R-2487) on fecal level will also be measured.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-75 years (Inclusive).
* Able to provide written informed consent.
* Men or women (not nursing or pregnant) who have active RA, defined as symptoms of RA prior to screening and have satisfied the ACR/EULAR 2010 criteria for the classification of RA prior to signing the informed consent.
* Subjects must have a CDAI > 10.0 at screening and have at least 3 tender and at least 3 swollen joints (excluding distal interphalangeal) at screening and at Day 1, based on the DAS28 joint count.
* Subjects may be able to be on hydroxychloroquine, methotrexate, and leflunomide. Sulfasalazine use is not permitted.
* Subjects may have received targeted synthetic DMARDs such as tofacitinib, baricitinib, and investigational therapies for RA if they have been washed out for 1 month prior to screening.
* Subjects receiving oral corticosteroids must be on a stable dose and at the equivalent of ≤10 mg prednisone daily for at least 4 weeks. Subjects may not receive an IM, IV or IA administration of a corticosteroid within 4 weeks prior to screening visit or initiation of therapy.
* All male and female subjects who are biologically capable of having children must agree to use a medically acceptable method of birth control for the duration of the study. All female subjects who are biologically capable of having children must have a negative pregnancy test result before administration of study drug. Any pregnancy that occurs in the female partner of a male subject in the trial must be reported if it occurs at any time during the study.
* Refrain from receiving any type of vaccinations during the study period (to include but not limited to influenza, COVID, shingles, tetanus, hepatitis, pneumonia, HPV, DPT, MMR, and polio).

Exclusion Criteria:

* Pregnancy (females, unless surgically sterile or at least two years post- menopausal must have a negative serum pregnancy test within 14 days prior to receiving the study drug and a negative urine pregnancy test on Study Day 0 before receiving the study drug).
* Nursing mothers.
* Subjects with autoimmune disease other than RA [e.g., psoriasis, systemic lupus erythematosus (SLE), vasculitis, seronegative spondylarthritis, Inflammatory Bowel Disease, Sjogren's syndrome] or currently active fibromyalgia.
* Subjects should not receive any of the following medications:
* Rituximab within 12 months prior to Day 1,
* Abatacept within 3 months prior to Day 1,
* Infliximab, Adalimumab, Certolizumab, Tocilizumab, Cyclosporine, or
* Mycophenolate mofetil within 2 months prior to Day 1, or
* Etanercept, Anakinra, Immunoglobulin, or blood products within 28 days prior to Day 1
* Prior immunotherapy, including systemic corticosteroids, such prednisone, biologics, Janus kinase (JAK) inhibitors (such as tofacitinib, baricitinib or upadacitinib), ozanimod, or investigational therapy must have completed at least 5 half-lives or 30 days, whichever is longer, prior to Day 0, unless otherwise specified. In the case of cell-depleting therapies, such as B or T cell depletion, cell counts must have recovered to acceptable or baseline levels (use of licensed agents for indications not listed in the package insert is permitted).
* Prior history of or current inflammatory joint disease other than RA (such as psoriatic arthritis, gout, reactive arthritis, Lyme disease).
* Subjects at risk for tuberculosis (TB) defined as follows: Current clinical, radiographic or laboratory evidence of active TB. Chest x-rays (posterior, anterior and lateral) obtained within the 3 months prior to obtaining written informed consent will be permitted but the images must be available and reviewed by the investigator. TB testing (IFN-gamma release assay or PPD) performed in the past month prior to Screening will be accepted; however, a copy of the report must be placed in the subject binder.
* A history of active TB.
* Subjects with a positive TB screening test indicative of latent TB including subjects currently being treated for latent tuberculosis infection (LTBI) will not be eligible for the study.
* Subjects with recent acute infection defined as:
* Any acute infection within 60 days prior to randomization that required hospitalization or treatment with parenteral antibiotics,
* Any acute infection within 30 days prior to randomization that required oral antimicrobial or antiviral therapy,
* Subjects with history of chronic or recurrent bacterial infection (such as chronic pyelonephritis, osteomyelitis, and bronchiectasis etc.),
* Subjects with any history of infection of a joint prosthesis or artificial joint,
* Subjects who have a history of systemic fungal infections (such as histoplasmosis, blastomycosis, or coccidiomycosis),
* Subjects with history of recurrent herpes zoster (more than 1 episode) or disseminated (more than 1 dermatome) herpes zoster or disseminated herpes simplex, or ophthalmic zoster will be excluded,
* Symptoms of herpes zoster or herpes simplex must have resolved more than 60 days prior to screening,
* Subjects with history of primary immunodeficiency.
* Subjects with history of Human Immunodeficiency Virus (HIV) infection or who tested positive for HIV.
* Evidence of infection with hepatitis B virus (HBV), hepatitis C virus (C), human immunodeficiency virus (HIV)-1 or HIV-2, or active infection with hepatitis A, as determined by results of testing at screening.
* Subjects who have a present malignancy or previous malignancy within the last 5 years prior to screening (except documented history of cured non- metastatic squamous or basal cell skin carcinoma or cervical carcinoma in situ). Subjects who had a screening procedure that is suspicious for malignancy, and in whom the possibility of malignancy cannot be reasonably excluded following additional clinical, laboratory or other diagnostic evaluations.
* Current clinical findings of a history of a demyelinating disorder.
* New York Heart Association (NYHA) Class III or IV heart failure.
* Subjects who have undergone a major surgical procedure within the 60 days prior to enrollment.
* Subjects for whom 5 or more joints cannot be assessed for tenderness or swelling (i.e. due to surgery, fusion, amputation, etc.).
* Current clinical findings of severe, progressive, or uncontrolled renal, hepatic, hematological, gastrointestinal, pulmonary, cardiac, endocrine, neurological, or cerebral disease with laboratory values as following:
* Hemoglobin level < 9.0 g/dL,
* Absolute white blood cell (WBC) count of <3.0×109/L (<3000/mm3), or absolute neutrophil count of <1.2×109/L (<1200/mm3), or absolute lymphocyte count of <0.8×109/L (<800/mm3),
* Thrombocytopenia, defined by platelet count <100×109/L (<100,000/mm3),
* Chronic kidney disease defined as Estimated glomerular filtration rate (eGFR) <60 mL/min/1.73m2, based on the age-appropriate calculation,
* Proteinuria ≥3+,
* Total bilirubin (T-bili), aspartate aminotransferase (AST), alanine aminotransferase (ALT) more than 1.5 times upper limit of normal (ULN)
* Previously diagnosed hepatic cirrhosis (Child Pugh A or higher) or previously diagnosed significant liver fibrosis (> F3).
* Any form of vaccination in the last 30 days, to include but not limited to influenza, COVID, shingles, tetanus, hepatitis, pneumonia, HPV, DPT, MMR, and polio.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Estimated)
Dates: Start 2023-10-19 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events and their relationship to R-2487 (probiotic) administration | Baseline through week 4
  To assess the number of participants with treatment-related adverse events after taking R-2487 (probiotic)

SECONDARY OUTCOMES:
Change in Disease Activity Score-28 Joint C-Reactive Protein (DAS28-CRP) | Baseline through week 4
  Change from Baseline in Disease Activity Score-28 joint C- Reactive Protein (DAS28-CRP) Score at Week 6 Describes severity of rheumatoid arthritis using clinical and laboratory data in swollen and tender joints. A score between 0 to 10 with the higher number indicating more active disease.
Change in Simplified Disease Activity Index (SDAI) Score over time | Baseline through week 4
  Baseline Simplified Disease Activity Index (SDAI) Score over time. The Simplified Disease Activity Index (SDAI) is the numerical sum of five outcome parameters: tender and swollen joint count (based on a 28-joint assessment), patient and physician global assessment of disease activity [visual analogue scale (VAS) 0-10 cm] and level of C-reactive protein (mg/dl, normal <1 mg/dl).

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - University of California, San Diego, San Diego, California
  - St.Jude Clinical Research, Doral, Florida
  - AP Medical Research, Miami, Florida
  - Altoona Center for Research, Duncansville, Pennsylvania
  - Prolato Clinical Research Center, Houston, Texas